CLINICAL TRIAL: NCT03439189
Title: Companion Protocol for the ¹³C-Methacetin Breath Test Using the BreathID® MCS System for Conatus Phase 2 Study of Emricasan, an Oral Caspase Inhibitor, Under Protocol IDN-6556-14 (NCT02960204)
Brief Title: Companion Protocol for Methacetin Breath Test (MBT) in Conatus Protocol IDN-6556-14
Status: Completed | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Collaborators: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CON-EX-0616
Record Dates: First submitted 2018-01-29; First posted 2018-02-20 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Hypertension, Portal | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Intervention Model Description: The population performing the MBT at weeks 24 and 48 will have approximately an equal number of subjects from each of the 4 parallel treatment arms (5 mg, 25 mg, 50 mg or placebo).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The collaborator is responsible for the masking process.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (4):
- Emricasan 5mg (Experimental): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (5 mg) twice a day. The MBT will be performed at screening, at week 24/week 48/at early termination.
  Interventions: Combination Product: Methacetin Breath Test; Drug: Emricasan
- Emricasan 25mg (Experimental): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (25 mg) twice a day. The MBT will be performed at screening, at week 24/ week 48/ at early termination.
  Interventions: Combination Product: Methacetin Breath Test; Drug: Emricasan
- Emricasan 50mg (Experimental): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (50 mg) twice a day. The MBT will be performed at screening, at week 24/ week 48/ at early termination.
  Interventions: Combination Product: Methacetin Breath Test; Drug: Emricasan
- Placebo (Placebo Comparator): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with a matching placebo twice a day. The MBT will be performed at screening, at week 24/week 48/at early termination.
  Interventions: Combination Product: Methacetin Breath Test; Drug: Placebo oral capsule

INTERVENTIONS:
Combination Product: Methacetin Breath Test — A breath analyzer will be used to measure changes in carbon-12 to carbon-13 ratio as a result of metabolism of the Methacetin substrate before and after treatment.
Drug: Emricasan — Investigational drug for NASH treatment in Main Conatus protocol
  Arms: Emricasan 25mg; Emricasan 50mg; Emricasan 5mg
Drug: Placebo oral capsule — Placebo versus emricasan in Conatus NASH treatment trial
  Arms: Placebo

SUMMARY:
To validate the ability of the Methacetin Breath Test (MBT) to detect clinically significant portal hypertension (CSPH)/severe portal hypertension (SPH) defined as hepatic venous pressure gradient (HVPG) ≥ 10 mmHg and HVPG ≥ 12 mmHg respectively, in patients with non-alcoholic steatohepatitis (NASH) during the course of treatment with Conatus's investigational product emricasan/placebo.

DETAILED DESCRIPTION:
This study is a companion protocol that will use the data generated by Conatus' study of emricasan under protocol IDN-6556-14 (NCT02960204).The IDN-6556-14 study is a Phase 2, multicenter, double-blind, randomized, placebo-controlled trial in subjects with non-alcoholic steatohepatitis (NASH) cirrhosis and severe portal hypertension.

As one of the Conatus' study exploratory objectives, this companion protocol is designed to assess whether emricasan compared to placebo improves liver metabolic function at Weeks 24 and 48 as assessed by the methacetin breath test (at select sites), if relevant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years or older, able to provide written informed consent and able to understand and willing to comply with the requirements of the study.
2. Cirrhosis due to NASH with exclusion of other causes of cirrhosis (e.g. chronic viral hepatitis, alcoholic liver disease, etc.)
3. Compensated cirrhosis OR Decompensated cirrhosis with no more than 1 prior significant decompensating event.
4. Severe portal hypertension defined as HVPG ≥12 mmHg
5. Subjects who are on NSBB, nitrates, diuretics, lactulose, rifaximin, or statins must be on a stable dose for at least 3 months prior to Day 1
6. Willingness to utilize effective contraception (for both males and females of childbearing potential) from Screening to 4 weeks after the last dose of study drug

Exclusion Criteria:

1. Evidence of severe decompensation
2. Severe hepatic impairment defined as a Child-Pugh score ≥10
3. ALT >3 times upper limit of normal (ULN) or AST >5 times ULN during screening
4. Estimated creatinine clearance <30 mL/min
5. Prior transjugular intrahepatic portosystemic shunt or other porto-systemic bypass procedure
6. Known portal vein thrombosis
7. Symptoms of biliary colic, e.g. due to symptomatic gallstones, within the last 6 months, unless resolved following cholecystectomy, other definitive treatment (e.g. sphincterotomy), or medical management (e.g. ursodeoxycholic acid)
8. Current use of medications that are considered inhibitors of OATP1B1 and OATP1B3 transporters
9. Alpha-fetoprotein >50 ng/mL
10. History or presence of clinically concerning cardiac arrhythmias, or prolongation of screening (pre-treatment) QTcF interval of >500 msec
11. History of or active malignancies, other than those successfully treated with curative intent and believed to be cured
12. Prior liver transplant
13. Change in diabetes medications or vitamin E within 3 months of screening
14. Uncontrolled diabetes mellitus (HbA1c >9%) within 3 months of screening
15. Significant systemic or major illness other than liver disease
16. HIV infection
17. Use of controlled substances (including inhaled or injected drugs) or non-prescribed use of prescription drugs within 1 year of screening
18. If female: planned or known pregnancy, positive urine or serum pregnancy test, or lactating/breastfeeding
19. Previous treatment with emricasan or active investigational medication (except methacetin) in a clinical trial within 3 months prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2016-08-28 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects that met the companion protocol eligibility criteria were enrolled.
Pre-assignment Details: Diagnostic endpoints used screening measurements taken prior to study drug administration, therefore no treatment effect was relevant. In addition, for the event prediction endpoints, the treatment covariate was tested for significance, and was found to be non-significant, thus removed from the final predicting model. As such, arms were combined.
Groups:
- ACLD With NASH: Subjects with advanced chronic liver disease (ACLD) and confirmed nonalcoholic steatohepatitis (NASH)
Period: Overall Study
Arm/Group | ACLD With NASH
Started | 343 (Subjects performed at least one Methacetin Breath Test (MBT))
Completed | 261
Not Completed | 82
Not completed — Protocol Violation | 19
Not completed — Lack of Efficacy | 63

BASELINE CHARACTERISTICS:
Population: Diagnostic endpoints used screening measurements taken prior to study drug administration, therefore no treatment effect was relevant. In addition, for the event prediction endpoints, the treatment covariate was tested for significance, and was found to be non-significant, thus removed from the final predicting model. As such, arms were combined.
Arm/Group | ACLD With NASH
Number analyzed (Participants) | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80
  Not Hispanic or Latino | 255
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 316
  More than one race | 2
  Unknown or Not Reported | 15
Region of Enrollment [Number; unit: participants]
  United States | 309
  France | 10
  Spain | 24
BMI [Mean (Standard Deviation); unit: kg/cm^2] | 35.3 (7.07)
Compensated (Liver disease) [Count of Participants; unit: Participants] | 265

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Matched Clinically Significant Portal Hypertension Based on Hepatic Venous Pressure Gradient (HVPG) and Methacetin Breath Test (MBT)
Description: Binary diagnosis of clinically significant portal hypertension (CSPH) as determined by HVPG, defined as HVPG ≥ 10mmHg and by the MBT derived from an algorithm developed under other Exalenz clinical studies
Time Frame: 1 hour for MBT related to assessment of this diagnostic primary outcome assesses during screening
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With CSPH: Subjects with Hepatic Venous Pressure Gradient (HVPG) equal to or greater than 10 mmHg
Arm/Group | Subjects With CSPH
Number analyzed (Participants) | 261
Participants | 190

2. Secondary Outcome: Number of Matched Subjects With Significant Portal Hypertension (Defined as HVPG>=12mmHg) Based on HVPG and MBT
Description: Binary diagnosis of HVPG>=12mmHg and by the MBT derived from an algorithm developed under other Exalenz clinical studies
Time Frame: 1 hour for MBT for assessment of this diagnostic secondary outcome assessed during screening
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Number of Subjects With SPH: Number of matched subjects with Severe Portal Hypertension (defined as HVPG>=12mmHg) based on HVPG and MBT.
Arm/Group | Number of Subjects With SPH
Number analyzed (Participants) | 261
Participants | 182

ADVERSE EVENTS:
Time Frame: Data was collected for a duration of approximately 1 year to observe the effect of the treatment. Additional MBTs after 24 and 48 weeks were performed to enable Conatus to assess the ability of MBT to identify improvement in liver function due to treatment, if relevant. Each MBT duration is 1 hour. The subsequent MBTs were not relevant to companion protocol primary and secondary efficacy diagnostic endpoints listed above, but additional safety information regarding these MBTs was collected.
Description: Diagnostic endpoints used screening measurements taken prior to study drug administration, therefore no treatment effect was relevant. In addition, for the event prediction endpoints, the treatment covariate was tested for significance, and was found to be non-significant, thus removed from the final predicting model. As such, arms were combined.
Arm/Group | ACLD With NASH
All-Cause Mortality (participants affected / at risk) | 0/343
Serious Adverse Events (participants affected / at risk) | 0/343
Other Adverse Events (participants affected / at risk) | 2/343
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACLD With NASH (N=343)
Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) — Cramps in the hands. (recorded as possibly related but occurred more than a month after MBT, so unlikely to be related.)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03439189/Prot_SAP_000.pdf